CLINICAL TRIAL: NCT01559064
Title: A Prospective, Observational Study of the Volumizing Effect of Open-Label Aesthetic Use of VOLUMA® in the Mid-Face Area
Brief Title: The Volumizing Effect of Juvéderm VOLUMA® in the Mid-Face
Status: Completed | Type: Observational
Sponsor: Allergan Medical (Industry)
Responsible Party: Sponsor
Organization: Allergan (Industry)
Other Study IDs: MAF/AGN/MED/FIL/017
Record Dates: First submitted 2012-03-19; First posted 2012-03-21 (Estimated); Results first posted 2013-06-10 (Estimated); Last update posted 2014-10-13 (Estimated); Status verified 2014-06

CONDITIONS: Age-related Volume Deficit in the Mid-face

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Age group A: Subjects 30 to 40 years old
  Interventions: Device: Crosslinked hyaluronic acid gel (Juvéderm VOLUMA®)
- Age group B: Subjects 40 to 50 years old
  Interventions: Device: Crosslinked hyaluronic acid gel (Juvéderm VOLUMA®)
- Age group C: Subjects over 50 years old
  Interventions: Device: Crosslinked hyaluronic acid gel (Juvéderm VOLUMA®)

INTERVENTIONS:
Device: Crosslinked hyaluronic acid gel (Juvéderm VOLUMA®) — All treatment details are at the discretion of the investigator and should be guided by the appropriate directions for use.
  Other Names: Juvéderm VOLUMA® with lidocaine

SUMMARY:
This is a prospective, observational study of the volumizing effect of aesthetic use of Juvéderm VOLUMA® with lidocaine in the mid-face area.

ELIGIBILITY:
Inclusion Criteria:

* Desire and willingness for correction of asymmetry or enhancement of his/her mid-face area.
* Be willing to undergo treatment for volume loss in the face area
* Females and males ≥30 years of age
* Be in good health as of the opinion of the Investigator
* Sign the Informed Consent Form prior to any study-related procedures being performed
* Have established a realistic treatment goal that the Investigator agrees is achievable i.e., have realistic expectations of aesthetic results

Exclusion Criteria:

* Have extensive tissue damage that could affect the aesthetic outcome
* Have a known allergy to any component of VOLUMA® with lidocaine injections
* Have an abscess or infection at the time of treatment that in the opinion of the Investigator does not make the subject eligible for the procedure.
* Have undergone cosmetic facial [e.g., face-lift, or other surgeries, which may alter the appearance of the mid-face region (laser, photomodulation intense pulsed light, radio frequency, dermabrasion, moderate or greater depth chemical peel, or other ablative procedures), tissue augmentation with dermal fillers or fat injections, or meso-therapy] anywhere in the mid-face region, or Botox® Cosmetic injections in the lower face (below the orbital rim), within the 6 months prior to entry in the study or be planning to undergo any of these procedures at any time during the study. NOTE: Prior treatment with hyaluronic acid (HA) fillers and/or collagen is allowed, provided the treatment was administered more than 6 months prior to study entry
* Have ever received semi-permanent fillers or permanent facial implants, e.g., calcium hydroxyapatite, L-polylactic acid, polymethylmethacrylate (PMMA), silicone, expanded polytetrafluoroethylene (ePTFE) anywhere in the lips, or be planning to be implanted with any of these products at any time during the study
* Have a history of anaphylaxis, multiple severe allergies, atopy, allergy to lidocaine (or any amide-based anesthetics), HA products, or Streptococcal protein, or be planning to undergo a desensitization therapy during the term of the study
* Suffer from an uncontrolled personality disorder (e.g., body dysmorphia, depression)
* Have a history of or currently suffer from an autoimmune disease (e.g., Rheumatoid arthritis, Crohn's disease)
* Have a history of streptococcal disease (e.g., strep throat or rheumatic fever with or without heart complications)
* Have a history of skin cancer
* Suffer from Porphyria
* Have epilepsy which is not controlled by anti-epilepsy therapy
* Current cutaneous inflammatory and/or infectious processes (e.g., acne, herpes, etc.)
* Have a history of treatment with interferon therapy (e.g., warfarin) or have taken non-steroidal anti-inflammatory drugs (NSAIDs) (e.g., aspirin, ibuprofen) or other substances known to increase coagulation time (e.g., herbal supplements with garlic or ginko biloba) within 10 days of undergoing study device injection. NOTE: Study device injection may be delayed as necessary to accommodate this 10-day washout period
* Be on a concurrent regimen of high doses of lidocaine (more than 400 mg) which may cause acute toxic reactions
* Be on a concurrent regimen of other local anesthetics structurally related to amide-type local anesthetics
* Have impaired cardiac conduction, severly impaired hepatic function, or severe renal dysfunction
* Have a condition or be in a situation that, in the Investigator's opinion, may put the subject at significant risk, may confound the study results, or may interfere significantly with the subject's participation in the study

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Normal, healthy subjects desiring aesthetic improvement
Sampling Method: Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2012-02; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Allergan Medical
Locations (4):
- Aalst, Belgium
- Cologne, North Rhine-Westphalia, Germany
- Naarden, Netherlands
- Mere Green, United Kingdom

REFERENCES:
- [Result] Philipp-Dormston WG, Eccleston D, De Boulle K, Hilton S, van den Elzen H, Nathan M. A prospective, observational study of the volumizing effect of open-label aesthetic use of Juvederm(R) VOLUMA(R) with Lidocaine in mid-face area. J Cosmet Laser Ther. 2014 Aug;16(4):171-9. doi: 10.3109/14764172.2014.910079. Epub 2014 May 5. PMID 24689357

RESULTS

PARTICIPANT FLOW:
Groups:
- Age Group A: Subjects 30 to 40 years old
  Crosslinked hyaluronic acid gel (Juvéderm VOLUMA®) : All treatment details are at the discretion of the investigator and should be guided by the appropriate directions for use.
- Age Group B: Subjects 40 to 50 years old
  Crosslinked hyaluronic acid gel (Juvéderm VOLUMA®) : All treatment details are at the discretion of the investigator and should be guided by the appropriate directions for use.
- Age Group C: Subjects over 50 years old
  Crosslinked hyaluronic acid gel (Juvéderm VOLUMA®) : All treatment details are at the discretion of the investigator and should be guided by the appropriate directions for use.
Period: Overall Study
Arm/Group | Age Group A | Age Group B | Age Group C
Started | 16 | 40 | 59
Completed | 15 | 39 | 57
Not Completed | 1 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Age Group A | Age Group B | Age Group C | Total
Number analyzed (Participants) | 16 | 40 | 59 | 115
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 16 | 40 | 50 | 106
  >=65 years | 0 | 0 | 9 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.7 (3.3) | 45.2 (2.8) | 58.3 (5.8) | 50.6 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 34 | 46 | 92
  Male | 4 | 6 | 13 | 23
Region of Enrollment [Number; unit: participants]
  Belgium | 0 | 4 | 6 | 10
  Netherlands | 3 | 4 | 13 | 20
  Germany | 8 | 25 | 33 | 66
  United Kingdom | 5 | 7 | 7 | 19

OUTCOME MEASURES:

1. Primary Outcome: Subject Experience Measured by Patient Satisfaction Questionnaire
Description: Subject satisfaction with treatment, based on a 5-point scale: (1) Delighted, (2) Happy, (3) Neutral, (4) Unhappy, (5) Very Unhappy
Time Frame: 3 weeks
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Age Group A | Age Group B | Age Group C
Number analyzed (Participants) | 16 | 39 | 57
Units on a scale | 1.94 (.68) | 1.62 (.78) | 1.51 (.57)

ADVERSE EVENTS:
Arm/Group | Age Group A | Age Group B | Age Group C
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/39 | 0/57
Other Adverse Events (participants affected / at risk) | 2/16 | 1/39 | 2/57
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Age Group A (N=16) | Age Group B (N=39) | Age Group C (N=57)
Injection site hematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Injection site edema (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Injection site pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Swelling (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No